CLINICAL TRIAL: NCT06077461
Title: The Effect of Mandala Coloring on Perceived Stress and Anxiety Levels in Type-2 Diabetes Patients: Randomized Controlled Study
Brief Title: The Effect of Mandala Coloring in Type-2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/ 12 - 41
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Mandala Painting; Type-2 Diabetic Patients

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:mandala painting (Experimental): Patients in this group will be subjected to mandala painting.
  Interventions: Behavioral: mandala painting
- Control (No Intervention): Patients in this group will not be subjected to mandala painting.

INTERVENTIONS:
Behavioral: mandala painting — Patients in this group will be subjected to mandala painting.
  Arms: Experimental:mandala painting

SUMMARY:
THIS RESEARCH was planned to examine the effect of mandala painting on the perceived stress and anxiety levels of type-2 diabetic patients.

DETAILED DESCRIPTION:
Diabetes is a frequently encountered chronic metabolic disease characterized by increased plasma glucose levels as a result of inadequate insulin secretion and/or increased insulin resistance. The most common type of diabetes is type-2 diabetes, accounting for approximately 90% of all cases. Type 2 diabetes is more common in middle and older ages, but today it is also seen in children and young adults due to negative changes in lifestyle habits.

Diabetes is typically a manageable disease through lifestyle changes and treatment. However, diabetes care can create additional stress for people with diabetes due to the never-ending demands of maintaining nutritional and physical health, exercising, monitoring blood sugar, regular monitoring, and managing fears about the reality of symptoms and complications. As a result, they experience feelings of depression, anxiety, and stress, which affects their health and overall quality of life. Patients with diabetes have significantly higher levels of anxiety and depression than the general population. The coexistence of diabetes and anxiety and stress results in poor glycemic control and self-management, increases the risk of diabetes complications, and reduces overall quality of life and life expectancy. Therefore, prevention, early recognition and treatment of these conditions are necessary to achieve optimal goals in the management and overall quality of life of patients.

A holistic approach should be adopted when planning the care practices of patients during this difficult period, and non-pharmacological practices should be planned, especially those that will allow the patient to perform daily life activities with minimum energy and maximum function. Mandala painting, one of the non-pharmacological practices, is an art therapy technique that can provide psychological support and healing. This circular art has traditionally been used for meditation in various Eastern cultures and is a symbol of psychological wholeness. Mandala coloring is a safe and accessible activity that does not require any special skills and can be used as a complementary strategy to support mental health. It is stated in the literature that painting mandalas improves psychological symptoms and relaxes the person. The artistic perspective of nursing is to understand the individual's needs, sources of worry, anxiety and stress, and then to develop practices that will increase his self-confidence and resilience by increasing his level of capability and competence. For this reason, this study was planned to examine the effect of mandala painting on the perceived stress and anxiety levels of Type-2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65

  * Having been diagnosed with Type-2 diabetes for at least 6 months
  * Being an inpatient in the endocrine clinic for at least 7 days
  * Not having a physical problem that would prevent painting mandalas (vision, hearing, etc.)

Exclusion Criteria:

* Not being able to use his hands actively
* Having a communication problem
* Having a learning problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | after 7 days
  The Perceived Stress Scale was developed by Cohen, Kamarck and Mermelstein in 1983 to determine the level of stress that threatens human health. Turkish validity and reliability were determined by Eskin et al. (2013). The scale is a 5-point Likert type scale and consists of 14 items. As the scores obtained from the scale increase, the level of stress perceived by the person also increases. PSS scores vary between 0 and 56, with 0-35 points indicating normal stress level and 35-56 points indicating that the individual is under stress.
State-Trait Anxiety Scale | after 7 days
  The State-Trait Anxiety Scale was developed by Spielberger et al. (1970). The validity and reliability of the scale in Turkey was determined by Öner and Le Compte (1983). The scale consists of two parts: State Anxiety Scale and Trait Anxiety Scale. The first 20 items evaluate situational anxiety, and the last 20 items evaluate trait anxiety. In this study, the scores obtained from the Scale, which is the first 20 items to evaluate situation-related anxiety, range between 20 and 80. Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No